CLINICAL TRIAL: NCT07034846
Title: Investigation of the Effects of Respiratory Muscle Training Combined With Otago Exercises in Elderly Patients Undergoing Coronary Artery Bypass Graft Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sadık Emre ÇELEBİ, MSc, PhD(c), Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/186
Record Dates: First submitted 2025-05-23; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Bypass Graft (CABG)
Keywords: Exercise; Inspiratory muscle training; Otago Exercises
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity intermittent IMT and Otago Exercises Group (Experimental): Patients aged 65 years and over who have undergone CABG surgery and who are at least 2 weeks postoperatively and who meet the inclusion criteria will be identified. Then, patients who volunteer to participate in the study will be referred.
  Interventions: Other: High-intensity intermittent IMT and Otago Exercises Group
- Sham IMT and Otago Exercises Group (Active Comparator): Patients aged 65 years and over who have undergone CABG surgery and who are at least 2 weeks postoperatively and who meet the inclusion criteria will be identified. Then, patients who volunteer to participate in the study will be referred.
  Interventions: Other: Sham IMT and Otago Exercises Group

INTERVENTIONS:
Other: High-intensity intermittent IMT and Otago Exercises Group — Patients in the experimental group will perform 7 sets of high-intensity intermittent inspiratory muscle training (IMT) for eight weeks, one day a week face-to-face with the researcher and two days at home, for a total of three days, each set consisting of 2 minutes of loading and 1 minute of rest for a total of 21 minutes. The Otago exercise program will be conducted for eight weeks, two days a week home-based and one day face-to-face with the researcher. The Otago exercise program will be complemented with walking exercise every day of the week. The Otago exercise program is designed to be progressive. The protocol was created to increase the difficulty of training at four different levels and every 2 weeks. The Otago exercise program will be applied to both the experimental group and the control group in the same protocol.
  Other Names: High-intensity intermittent IMT group
  Arms: High-intensity intermittent IMT and Otago Exercises Group
Other: Sham IMT and Otago Exercises Group — Patients in the control group will perform 7 sets of sham inspiratory muscle training (IMT), consisting of 2 minutes of loading and 1 minute of rest in each set for a total of 21 minutes, one day a week face-to-face with the researcher and two days at home, for eight weeks. The Otago exercise program will be conducted for eight weeks, two days a week home-based and one day face-to-face with the researcher. The Otago exercise program will be complemented with walking exercise every day of the week. The Otago exercise program is designed to be progressive. The protocol was created to increase the difficulty of training at four different levels and every 2 weeks. The Otago exercise program will be applied to both the experimental group and the control group in the same protocol.
  Other Names: Sham IMT group
  Arms: Sham IMT and Otago Exercises Group

SUMMARY:
A review of the literature suggests that high-intensity intermittent inspiratory muscle training (IMT) combined with the Otago exercise program may provide positive effects on early post-discharge recovery of patients aged 65 years and older undergoing coronary artery bypass graft (CABG) surgery. No studies have yet examined the effects of high-intensity intermittent IMT combined with the Otago exercise program on patients undergoing CABG surgery. This study is the first to evaluate the effects of high-intensity intermittent IMT combined with the Otago exercise program on pulmonary function, functional capacity, muscle strength, functional mobility, balance, anxiety and depression levels, frailty, and quality of life in elderly patients undergoing CABG surgery.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgery aims to revascularize the myocardium by bypassing one or more coronary arteries narrowed or occluded due to atherosclerosis. Procedures such as sternotomy, cardiopulmonary bypass, general anesthesia, and pleural drain placement can lead to postoperative complications including hypersecretion, hypoxemia, decreased pulmonary compliance, reduced exercise capacity, and impaired lung function. These complications may cause prolonged immobilization and additional pulmonary issues. Moreover, protein catabolism after cardiovascular surgery leads to muscle protein loss, which is exacerbated by immobilization, slowing protein synthesis and accelerating muscle fiber breakdown and cell death, thereby contributing to muscle loss progression. Postural balance also decreases following CABG, potentially leading to reduced functional activities, increased fall risk, morbidity, and mortality. CABG negatively impacts patients' quality of life and causes functional limitations. Anxiety about disease recurrence and fear of death after discharge contribute to psychological stress for patients and relatives, further impairing recovery.

Frailty is closely associated with cardiopulmonary diseases and is common after CABG surgery. A study evaluating 180 bypass patients with an average age of approximately 69 years found that 23.3% were frail. High frailty scores post-CABG correlate with adverse outcomes such as prolonged hospital stays and rehospitalization within 30 days.

Inspiratory muscle training (IMT) is a method designed to strengthen inspiratory muscles by providing airway resistance during breathing. Effective IMT requires appropriate intensity, duration, and frequency. Training at or above 30% of maximal inspiratory pressure (MIP) for 20-30 minutes daily, five days a week, over 5-12 weeks produces structural changes in respiratory muscles.

Previous studies demonstrated that IMT improves inspiratory muscle strength, functional capacity, psychosocial status, and quality of life in patients undergoing CABG surgery. Additionally, moderate to high-intensity IMT combined with aerobic and strengthening exercises during cardiac rehabilitation increases exercise capacity, inspiratory muscle strength, and quality of life more than sham IMT combined with similar exercises.

High-intensity intermittent IMT has recently shown beneficial results in cardiovascular and pulmonary diseases. In heart failure patients, high-intensity intermittent IMT performed in cycles of loading and rest improved dyspnea, frailty, fatigue, inspiratory muscle strength, respiratory muscle endurance, exercise capacity, and quality of life, compared to sham IMT. Similar positive effects were observed in patients with bronchiectasis and elderly individuals undergoing home-based IMT, with improvements in inspiratory muscle function, balance, and physical performance.

IMT has demonstrated effectiveness in reducing dyspnea, improving respiratory muscle strength, pulmonary function, functional capacity, daily living activities, and quality of life in patients with chronic obstructive pulmonary disease, chronic kidney disease, chronic heart failure, and in healthy populations. It also enhances postural stability due to the diaphragm's mechanical role in lumbar stabilization.

The Otago exercise program, developed in New Zealand to prevent falls, is a home-based training protocol including warm-up, strengthening, balance, and walking exercises. Performed three times weekly with progressively increasing intensity, it improves lower extremity muscle strength, balance, and mobility in elderly individuals.

Few studies have investigated the combination of IMT and the Otago exercise program. Recent research in healthy adults and diabetic patients indicates that combined training improves balance, inspiratory muscle function, mobility, respiratory function, muscle strength, and endurance more than either intervention alone.

This prospective, randomized, controlled, single-blind study will evaluate the effects of the Otago exercise program combined with high-intensity IMT on elderly patients undergoing CABG surgery. The study will be conducted at Istanbul University-Cerrahpaşa Cardiology Institute, Department of Cardiovascular Surgery.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older undergoing coronary artery bypass graft surgery
* Hospital discharge realized (post operative ≥ 2 weeks)
* No contraindications for exercise training
* Not concurrently participating in another exercise training program
* Have the means to enter a home-based rehabilitation program
* Patients who agree to participate voluntarily will be included in the study program.

Exclusion Criteria:

* Cardiovascular instability (aortic dissection, unstable angina pectoris, acute decompensated heart failure, acute pericarditis or myocarditis, severe cardiac arrhythmia, ventricular aneurysm)
* Uncontrolled hypertension and diabetes mellitus
* Diagnosed with chronic lung disease
* Cognitive impairment that prevents them from communicating with the physiotherapist
* Failure to maintain the exercise training program
* Patients with severe orthopedic or neurological disorders will not be included.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum inspiratory pressure | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  In the maximum inspiratory pressure measurement, patients will be asked to perform maximum inspiration for at least 2 seconds through the mouthpiece after first performing maximum expiration by sitting and using a nose clip. The measurement result will be recorded in units of cmH2O and percentage % of the expected value. The measurement will be considered satisfactory when a change of less than 10% is observed between the three measurements and the highest value is adopted.

SECONDARY OUTCOMES:
Maximum expiratory pressure | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Patients will be asked to perform maximum expiration against a closed system for at least 2 seconds after maximum inspiration. The measurement result will be recorded in units of cmH2O and percentage % of the expected value. The measurement will be considered satisfactory when a change of less than 10% is observed between the three measurements and the highest value is adopted.
Forced vital capacity (FVC) massessment | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Patients will perform a rapid and complete inhalation maneuver from functional residual capacity to total lung capacity, followed by a continuous and maximal exhalation maneuver lasting at least six seconds. Verbal and non-verbal encouragement will be provided throughout the maneuvers. The test will be terminated once acceptable repeatability is achieved. The results will be recorded in litres.
Assessment of functional capacity | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Functional capacity will be assessed using the 6-Minute Walk Test. Patients will be instructed to walk at their own pace to cover the maximum possible distance along a 30-meter corridor within 6 minutes. The total distance walked will be recorded in meters. Heart rate, measured in beats per minute, blood pressure, measured in millimeters of mercury, and oxygen saturation, measured as a percentage, will be recorded both before and after the test. Patients will be informed that they may rest or slow down as needed during the test.
Evaluation of muscle strength | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Isometric muscle strength of the M. Quadriceps femoris will be measured using a portable handheld dynamometer. Patients will be seated with the knee in full extension, and maximum resistance will be applied at the ankle to assess muscle strength. The measurement will be repeated three consecutive times, and the average value will be recorded in kilograms.
Assessment of functional mobility | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Mobility will be assessed using the Timed Up and Go Test. Patients will be instructed to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. The total time taken to complete this task will be recorded in seconds. A time of 13.5 seconds or longer is indicative of a higher risk of falls.
Balance assessment | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Balance performance will be assessed using the Berg Balance Scale, which consists of 14 items scored from 0 to 4, with a maximum total score of 56. Scores between 0-20 indicate balance impairment, 21-40 indicate acceptable balance, and 41-56 indicate good balance performance. Additionally, balance confidence will be evaluated using the Activity Specific Balance Confidence Scale, which includes 16 questions assessing confidence in performing daily activities indoors and outdoors. Each item is scored from 0% (unsafe) to 100% (completely safe), and the average score is calculated to provide an overall balance confidence percentage. Higher scores represent greater confidence.
Assessment of anxiety and depression level | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Anxiety and depression levels will be assessed using the Hospital Anxiety and Depression Scale. This scale evaluates the risk and severity of anxiety and depression symptoms through 14 questions-seven assessing anxiety (odd-numbered) and seven assessing depression (even-numbered). Responses are rated on a four-point Likert scale ranging from 0 to 3. The total score ranges from 0 to 42. Higher scores indicate more severe symptoms.
Frailty assessment | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Frailty will be assessed using the Fried Frailty Phenotype based on five criteria: Participants with three or more criteria will be classified as frail.
Assessment of quality of life | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Patients' quality of life will be assessed using the Short Form-36 questionnaire, which comprises 36 items covering eight subscales related to physical and mental health. Each subscale is scored between 0 and 100, with higher scores indicating a better overall quality of life.
Forced expiratory volume in one second (FEV1) assessment | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Patients will perform a rapid and complete inhalation maneuver from functional residual capacity to total lung capacity, followed by a continuous and maximal exhalation maneuver lasting at least six seconds. Verbal and non-verbal encouragement will be provided throughout the maneuvers. The test will be terminated once acceptable repeatability is achieved. The results will be recorded in litres.
FEV1/FVC ratio | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  FVC and FEV1 results will be compared and expressed as percentages.
Forced expiratory flow 25-75% (FEF25-75) assessment | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Patients will perform a rapid and complete inhalation maneuver from functional residual capacity to total lung capacity, followed by a continuous and maximal exhalation maneuver lasting at least six seconds. Verbal and non-verbal encouragement will be provided throughout the maneuvers. The test will be terminated once acceptable repeatability is achieved. The results will be expressed in litres per second.
Peak expiratory flow (PEF) assessment | The baseline assessment will be conducted at 2 weeks post-surgery. Following the completion of the 8-week intervention protocol, the final assessment will be performed at 10 weeks post-surgery.
  Patients will perform a rapid and complete inhalation maneuver from functional residual capacity to total lung capacity, followed by a continuous and maximal exhalation maneuver lasting at least six seconds. Verbal and non-verbal encouragement will be provided throughout the maneuvers. The test will be terminated once acceptable repeatability is achieved. The results will be expressed in litres per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Rengin Demir, Professor, Study Director — Istanbul University-Cerrahpaşa, Cardiology Institute, Department of Cardiology
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including all measurement data collected in the study, will be shared with researchers upon request. The data will become available after the completion of the study and publication of the results, and will remain accessible for 5 years thereafter. Researchers may request access via email at celebisaemre@gmail.com. No formal approval process will be required to obtain the data.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be available beginning in June 2025 and will remain accessible through June 2030.
Access Criteria: Access to de-identified individual participant data (IPD) and supporting information will be available to qualified researchers upon request. Researchers interested in accessing the data may contact via email at celebisaemre@gmail.com. There will be no requirement to submit a formal research proposal, data sharing agreement, or obtain prior approval. The data provided will include all measurement data collected in the study, de-identified to protect participant privacy.
  Requests will be handled on a first-come, first-served basis and no independent review or committee approval is necessary. The data may be used for secondary analyses, validation studies, or meta-analyses.